CLINICAL TRIAL: NCT01685216
Title: A Multi-center, Open-label, Efficacy and Safety Study of Velaglucerase Alfa Enzyme Replacement Therapy in Children and Adolescents With Type 3 Gaucher Disease
Brief Title: Efficacy and Safety Study of Velaglucerase Alfa in Children and Adolescents With Type 3 Gaucher Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGT-GCB-068; 2012-003427-38 (EudraCT Number)
Record Dates: First submitted 2012-09-10; First posted 2012-09-14 (Estimated); Results first posted 2015-10-30 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Gaucher Disease, Type 3
Keywords: VPRIV; velaglucerase alfa
MeSH Terms: conditions — Gaucher Disease | interventions — Glucosylceramidase; Enzyme Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- velaglucerase alfa (Experimental): IV infusion, 60 U/kg, every other week for 1 year
  Interventions: Biological: velaglucerase alfa

INTERVENTIONS:
Biological: velaglucerase alfa — lyophilized powder, intravenous infusion, units, Every other week (EOW)
  Other Names: VPRIV; Gene activated glucocerebrosidase; GA-GCB; Enzyme replacement therapy

SUMMARY:
Gaucher disease is a rare lysosomal storage disorder caused by the deficiency of the enzyme glucocerebrosidase (GCB). Gaucher disease has been classified into 3 clinical subtypes based on the presence or absence of neurological symptoms and the severity of these neurological symptoms. Patients with type 2 Gaucher disease present with acute neurological deterioration, and those with type 3 disease typically display a more sub acute neurological course. Type 1 Gaucher disease, the most common form accounting for more than 90% of all Gaucher disease cases, does not involve the central nervous system.

The purpose of this clinical research study is to investigate the safety and effectiveness of velaglucerase alfa in patients with type 3 Gaucher disease.

DETAILED DESCRIPTION:
Gaucher disease is a rare lysosomal storage disorder caused by the deficiency of the enzyme glucocerebrosidase (GCB). Due to the deficiency of functional GCB, glucocerebroside accumulates within the macrophages leading to cellular engorgement, organomegaly, and organ system dysfunction. Gaucher disease has been classified into 3 clinical subtypes based on the presence or absence of neurological symptoms and severity of neurological symptoms. Patients with type 2 Gaucher disease present with acute neurological deterioration, and those with type 3 Gaucher disease typically display a more sub acute neurological course; type 1 Gaucher disease, the most common form accounting for more than 90% of all cases, does not involve the central nervous system.

Velaglucerase alfa is an approved enzyme replacement therapy (ERT) for pediatric and adult patients with type 1 Gaucher disease. ERTs have been proven to reduce organomegaly, improve hematological parameters and positively impact health-related quality of life; ERTs have not been shown to cross the blood brain barrier and as a result have shown limited ability to improve the neurological (Central Nervous System; CNS) manifestations associated with Gaucher disease.

This study will provide a basis for exploring the efficacy and safety of velaglucerase alfa in patients with type 3 Gaucher disease.

ELIGIBILITY:
Inclusion Criteria: Each patient must meet the following criteria to be enrolled in this study.

1. The patient has a confirmed diagnosis of type 3 Gaucher disease.
2. The patient is ≥ 2 and < 18 years of age at the time of enrollment.
3. The patient is either näive to treatment or has not received treatment (investigational or approved) for Gaucher disease within 12 months prior to study entry.
4. The patient has Gaucher disease-related anemia, defined as hemoglobin concentration below the lower limit of normal for age and sex.

   AND ONE OR MORE OF THE FOLLOWING THREE CRITERIA
   * The patient has at least moderate splenomegaly (2 to 3 cm below the left costal margin) by palpation.
   * The patient has Gaucher disease-related thrombocytopenia, defined as platelet count < 120 x 10,000 platelets/cubic mm.
   * The patient has a Gaucher disease-related readily palpable enlarged liver.
5. Patients who have undergone splenectomy may still be eligible to participate in the study.
6. Female patients of child-bearing potential must agree to use a medically acceptable method of contraception at all times during the study. Pregnancy testing will be performed at the time of enrollment and as required throughout participation in the study. Male patients must agree to use a medically acceptable method of contraception at all times during the study and report a partner's pregnancy to the Investigator.
7. The patient's parent(s) or the patient's legally authorized representative(s) has provided written informed consent that has been approved by the Institutional Review Board/Independent Ethics Committee (IRB/IEC).

Exclusion Criteria: Patients who meet any of the following criteria will be excluded from this study.

1. The patient is suspected of having type 2 or type 1 Gaucher disease.
2. The patient is < 2 years of age.
3. The patient has experienced a severe (Grade 3 or higher) infusion-related hypersensitivity reaction (anaphylactic or anaphylactoid reaction) to any enzyme replacement therapy for Gaucher disease (approved or investigational).
4. The patient has received any non-Gaucher disease-related treatment with an investigational drug within 30 days prior to study entry.
5. The patient is a pregnant and/or lactating female.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2012-09-14 (Actual); Primary Completion 2015-03-15 (Actual); Study Completion 2015-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- Egypt (3):
  - Alexandria University Hospital, Alexandria
  - Abu El Rich Hospital, Cairo University Hospital, Cairo
  - Children's Hospital, Ain Shams University Hospital, Cairo
- KEM Hospital Research Centre, Pune, Maharashtra, India
- Hospital La Rabta, Tunis, Tunisia

RESULTS

PARTICIPANT FLOW:
Groups:
- Velaglucerase Alfa: Participants received an intravenous (IV) infusion of velaglucerase alfa at 60 U/kg, every other week for 1 year, then were followed for 1 month.
Period: Overall Study
Arm/Group | Velaglucerase Alfa
Started | 7
Completed | 6
Not Completed | 1
Not completed — Did not receive study drug | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat population, defined as all participants who received at least 1 study drug infusion (full or partial).
Arm/Group | Velaglucerase Alfa
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.17 (4.446)
Age, Customized [Count of Participants; unit: Participants]
  2 to 4 years | 4
  5 to 17 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 12 Months (Week 53) in Hemoglobin Concentration
Description: Hemoglobin concentration was measured as part of the hematology panel or measured separately when the hematology panel was not scheduled. Samples were measured by a central laboratory. Baseline is the modified baseline hemoglobin concentration, the average of the values from screening, baseline, and Week 1/Day 1. A positive change from baseline indicates that hemoglobin concentration increased.
Time Frame: Baseline, Week 53 or end of study
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Velaglucerase Alfa
Number analyzed (Participants) | 6
g/dL | 2.15 (1.213)

2. Secondary Outcome: Change From Baseline to 12 Months (Week 53) in Platelet Count
Description: Platelet count was measured at a central laboratory as part of the hematology panel. Baseline is the modified baseline platelet count, the average of the values from screening, baseline and Week 1/Day 1. A positive change from baseline indicates that platelet count increased.
Time Frame: Baseline, Week 53
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: platelets (x10^9)/L
Arm/Group | Velaglucerase Alfa
Number analyzed (Participants) | 6
platelets (x10^9)/L | 136.6 (51.48)

3. Secondary Outcome: Percent Change From Baseline to 12 Months (Week 51) in Normalized Liver Volume Measured Using Magnetic Resonance Imaging (MRI)
Description: Quantitative abdominal MRI was used to measure liver volume. If sedation was necessary to perform an MRI and the investigator deemed that this would be an unwarranted risk to the participant, liver volume could have been measured by ultrasound. Organ volume was measured by a single independent reviewer who was blinded to the participant identification and time point. The liver size relative to body weight was determined using the corresponding body weight measured at the same visit. Change in liver volume is presented as the normalized percentage of body weight. A negative change from baseline indicates that liver volume decreased.
Time Frame: Baseline, Week 51 or end of study
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Velaglucerase Alfa
Number analyzed (Participants) | 6
percent change | -30.12 (10.366)

4. Secondary Outcome: Percent Change From Baseline to 12 Months (Week 51) in Normalized Spleen Volume Measured Using Magnetic Resonance Imaging (MRI)
Description: Quantitative abdominal MRI was used to measure spleen volume. If sedation was necessary to perform an MRI and the investigator deemed that this would be an unwarranted risk to the participant, spleen volume could have been measured by ultrasound. Organ volume was measured by a single independent reviewer who was blinded to the participant identification and time point. The spleen size relative to body weight was determined using the corresponding body weight measured at the same visit. Change in spleen volume is presented as the normalized percentage of body weight. A negative change from baseline indicates that spleen volume decreased.
Time Frame: Baseline, Week 51
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Velaglucerase Alfa
Number analyzed (Participants) | 6
percent change | -62.27 (19.991)

5. Secondary Outcome: Number of Participants With Abnormal Neurological Status During The Study
Description: Neurological symptoms were evaluated at regular intervals during the study and assessed on an individualized basis by a limited, age- and developmental stage-appropriate neurological examination adapted to suit the status of each participant. It was preferred that each neurological examination be performed by a neurologist with experience in assessment of neurological symptoms in patients with Gaucher disease and, if possible, the same neurologist (or designee) who evaluated a given participant at baseline performed the neurological examinations scheduled for that participant during the treatment phase and at the end of study visit.
Time Frame: Baseline, Weeks 13, 25, 37, and 53 or end of study
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Velaglucerase Alfa
Number analyzed (Participants) | 6
participants | 6

6. Secondary Outcome: Number of Participants Who Experienced a Treatment-Emergent Adverse Event
Description: Adverse events (AEs) were monitored continuously throughout the study from the time the participant or participants parent/legal guardian signed the informed consent/assent (if applicable) until 30 days after the participant's last dose of study drug or at the end of study visit and/or until the event resolved or stabilized, or an outcome had been reached, whichever came first. Treatment-emergent adverse events (TEAEs) were defined as AEs which occurred on or after the time of the first infusion until 30 days after the participant's last study infusion. An infusion-related reaction is defined as an AE that 1) began either during or within 12 hours after the start of the infusion, and 2) was judged as possibly or probably related to study medication.
Time Frame: 57 weeks
Population: The Safety Analysis population, defined as all participants who received at least 1 study drug infusion (full or partial).
Measure: Number; unit: participants
Arm/Group | Velaglucerase Alfa
Number analyzed (Participants) | 6
participants
  Any TEAE | 6
  Serious TEAE | 1
  Infusion-related TEAE | 1

7. Secondary Outcome: Number of Participants Who Developed Anti-Velaglucerase Alfa Antibodies During The Study
Description: Participants provided blood samples for measurement of anti-velaglucerase alfa antibodies in serum at baseline and approximately every 12 weeks during the treatment phase. Blood samples collected during the treatment phase were to be drawn prior to infusions. Analysis of anti-velaglucerase antibodies used a validated 3-tier immunoassay method (screening, confirmatory, and titer).
Time Frame: Baseline, Weeks 13, 25, 37 and 53
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Velaglucerase Alfa
Number analyzed (Participants) | 6
participants
  Baseline | 0
  Week 13 | 1
  Week 25 | 1
  Week 37 | 1
  Week 53 | 1

ADVERSE EVENTS:
Description: Treatment-emergent adverse events are reported for the Safety population, defined as all participants who received at least 1 study drug infusion (full or partial).
Arm/Group | Velaglucerase Alfa
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Velaglucerase Alfa (N=6)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Velaglucerase Alfa (N=6)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Strabismus (Eye disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (5)
Gingival bleeding (Gastrointestinal disorders) | 1 (2)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 4 (17)
Gait disturbance (General disorders) | 1 (2)
Influenza like illness (General disorders) | 1 (2)
Asthenia (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 2 (4)
Acute tonsillitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Postprocedural cellulitis (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (8)
Convulsion (Nervous system disorders) | 1 (2)
Fine motor delay (Nervous system disorders) | 1 (1)
Gross motor delay (Nervous system disorders) | 1 (1)
Muscle spasticity (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Heat rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Chilblains (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.